CLINICAL TRIAL: NCT02278952
Title: Tacrolimus Adjustment by NFAT-related Gene Expression in Lung Allograft Recipients.
Acronym: TANGELA
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Astellas Scientific & Medical Affairs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Astellas ISR000990
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Transplantation, Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-interventional cohort study to assess a novel assay to detect excessive or insufficient immunosuppression from the drug tacrolimus in lung transplant recipients. The assay measures mean residual expression (MRE) of genes downstream of nuclear factor of activated T cells (NFAT), a transcription factor regulated by tacrolimus. The investigators will assess whether MRE levels identify subjects at risk for rejection (insufficient immunosuppression) or infection (excessive immunosuppression).

ELIGIBILITY:
Inclusion criteria:

The study will include lung allograft recipients within 2 months of transplantation at UCSF.

Exclusion criteria:

Subjects will be excluded who are (a) unable to provide consent or (b) if treating clinicians do not anticipate subject will start on tacrolimus. Recruitment and enrollment in this study are targeted equally between women and minorities and the study will not exclude any gender or racial/ethnic group. This study does not involve vulnerable populations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greenland John, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Lung transplant recipients treated at UCSF with tacrolimus-based immunosuppressive regimen recruited one to two months post-transplant.
Pre-assignment Details: Participants followed for 6 to 18 months post transplantation. Study visits performed within one day of a clinical bronchoscopy scheduled either for cause, such as suspected infection or rejection, or for surveillance at 2, 3, 6, 12, or 18 months.
Units Other Than Participants: Biopsies
Groups:
- Lung Transplant Participants: Lung transplant participants treated at UCSF with tacrolimus-based immunosuppression were followed until 18 months post-transplant, or until the participant's death or withdrawal.
Period: Overall Study
Arm/Group | Lung Transplant Participants
Started | 50; 225 Biopsies (The number of biopsy procedures performed during the time the patient was enrolled in the study.)
Completed | 44; 117 Biopsies (The number of biopsy samples assayed during the time the patient was enrolled in the study.)
Not Completed | 6; 108 Biopsies
Not completed — Insufficient Sample | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lung Transplant Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Lung Disease Diagnosis Group [Count of Participants; unit: Participants]
  A-Obstructive | 8
  B-Pulmonary vascular | 1
  C-Cystic Fibrosis | 2
  D-Restrictive | 33

OUTCOME MEASURES:

1. Primary Outcome: Association of Percentage of Mean Residual Expression (MRE%) of NFAT-related Cytokine Expression and Acute Cellular Rejection
Description: The prescribed tacrolimus dosage was determined by the treating physician who was not aware of the study-assay values. For the study assay, two blood draws were collected at a study visit during the assessment period (from 1 month up to 18 months post-transplant). The first draw occurred before tacrolimus dosage (trough) and the second occurred 90 to 120 minutes after tacrolimus dosage (peak). To determine MRE, whole blood was stimulated, RNA was extracted, and residual expression of NFAT-related cytokines (NFAT: nuclear factor of activated T-cells) was determined by quantitative polymerase chain reaction (qPCR). Researchers stratified blood draws based on subject's rejection pathology at time of blood draw and observed percentage distribution of MRE values within each rejection pathology group. Observed differences between MRE distributions within non-rejection group and rejection groups.
Time Frame: from 1 month up to 18 months post-transplant
Population: Number of participants' study visits analyzed determined by the availability and quality of samples at both time points.
Measure: Mean (Standard Error); unit: percentage of mean residual expression
Units Other Than Participants: biopsies
Groups:
- Non-rejection: Blood draw samples collected at the time of bronchoscopy with biopsy. Samples included if both time points (before tacrolimus dose and 90 to 120 minutes after dose) were collected, samples provided good quality RNA, and the patient had no evidence of acute cellular rejection. Acute cellular rejection was determined based on clinical interpretation of transbronchial biopsy specimens and graded according to International Society of Heart and Lung Transplantation (ISHLT) guidelines, with non-rejection defined as "A0B0."
- Rejection: Transbronchial biopsy showing A>0 or B>0 pathology with no rejection defined as A = 0 in perivascular interstitial components of the lung and B = 0 in airway components of the lung.
Arm/Group | Non-rejection | Rejection
Number analyzed (Participants) | 33 | 11
Number analyzed (biopsies) | 106 | 11
percentage of mean residual expression | 39.5 (2.9) | 41.7 (6.9)
Statistical Analysis 1: Comparison: Non-rejection vs Rejection; Test type: Other — Generalized estimating equation-adjusted linear models; p = 0.33, GEE-adjusted models

2. Primary Outcome: Association of Percentage of Mean Residual Expression (MRE%) of NFAT-related Cytokine Expression and Infection
Description: Researchers stratified blood draws based on subject's airway infection status at time of blood draw (based on biopsy results) and observed percentage distribution of MRE values within each infection status group. Researchers observed differences between MRE distributions within subjects with airway infection at time of blood draw and subjects with no infection diagnosis.
Time Frame: from 1 month up to 18 months post-transplant
Population: Number of participants' study visits
Measure: Mean (Standard Deviation); unit: percentage of mean residual expression
Units Other Than Participants: biopsies
Groups:
- Non-Infection: No airway infection as defined by presence of pathogenic species on bronchoalveolar lavage (BAL) culture and at least one of the following: semi-quantitative cultures with at least moderate quantity, CT findings, or symptoms consistent with acute infection.
- Infection: Airway infection defined by presence of pathogenic species on BAL culture and at least one of the following: semi-quantitative cultures with at least moderate quantity, CT findings, or symptoms consistent with acute infection.
Arm/Group | Non-Infection | Infection
Number analyzed (Participants) | 32 | 12
Number analyzed (biopsies) | 100 | 17
percentage of mean residual expression | 14.4 (2.9) | 22.2 (4.6)
Statistical Analysis 1: Comparison: Non-Infection vs Infection; Test type: Other — Generalized estimating equation-adjusted linear model; p < 0.0001, GEE-adjusted linear model

3. Secondary Outcome: Association of Percentage of Mean Residual Expression (MRE%) of NFAT-related Cytokine Expression and Weeks Post-Transplant
Description: Researchers observed percentage distribution of MRE values at time of blood draw from study visits at 4 weeks post-transplant up to 82 weeks post-transplant. Researchers observed association between percentage of MRE at time of blood draw and the number of weeks post-transplant.
Time Frame: from 1 month (4 weeks) up to 18 months (82 weeks) post-transplant
Population: Number of participants' study visits
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of mean residual expression
Units Other Than Participants: biopsies
Groups:
- Lung Transplant Participants: Time post-transplant determined by the number of weeks between the transplant date and the date of the blood draw. Outcome measures how mean residual expression values as a function of time post-transplant.
Arm/Group | Lung Transplant Participants
Number analyzed (Participants) | 44
Number analyzed (biopsies) | 117
percentage of mean residual expression | 0.35 [0.04 to 0.66]
Statistical Analysis 1: Comparison: Lung Transplant Participants; Test type: Other — Generalized estimating equation-adjusted linear models; p = 0.049, GEE-adjusted linear models

4. Secondary Outcome: Association of Percentage of Mean Residual Expression (MRE%) of NFAT-related Cytokine Expression and Tacrolimus Trough Level
Description: Researchers observed percentage distribution of MRE values on the day of blood draws. Researchers measured tacrolimus concentration in blood drawn before tacrolimus dosage (trough) and observed the association between percentage of MRE on the day of blood draw and tacrolimus trough level.
Time Frame: from 1 month up to 18 months post-transplant
Population: Number of participants' study visits
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of mean residual expression
Units Other Than Participants: biopsies
Groups:
- Lung Transplant Participants: Lung transplant participants treated at UCSF with tacrolimus-based immunosuppression were followed until 18 months post-transplant, or until the participant's death or withdrawal. Tacrolimus trough levels were assayed on whole blood by the clinical lab using the Architect Immunoassay. The tacrolimus trough value closest in time to the study visit used.
Arm/Group | Lung Transplant Participants
Number analyzed (Participants) | 44
Number analyzed (biopsies) | 117
percentage of mean residual expression | -1.687 [-3.714 to 0.397]
Statistical Analysis 1: Comparison: Lung Transplant Participants; Test type: Other — Generalized estimating equation-adjusted linear models; p = 0.114, GEE-adjusted linear models

5. Secondary Outcome: Association of Percentage of Mean Residual Expression (MRE%) of NFAT-related Cytokine Expression and Medication Dosages
Description: Researchers observed percentage distribution of MRE values on the day of blood draws and measured tacrolimus, prednisone, and mycophenolate dose at the time of blood draw. Researchers observed the association between percentage of MRE on the day of blood draw and tacrolimus, prednisone, and mycophenolate dose, respectively, at the time of blood draw.
Time Frame: from 1 month up to 18 months post-transplant
Population: Number of participants' study visits
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of mean residual expression
Units Other Than Participants: biopsies
Groups:
- Lung Transplant Participants: Lung transplant participants treated at UCSF with tacrolimus-based immunosuppression were followed until 18 months post-transplant, or until the participant's death or withdrawal. Tacrolimus, prednisone, and mycophenolate dose abstracted from medical charts at the time of blood draw.
Arm/Group | Lung Transplant Participants
Number analyzed (Participants) | 44
Number analyzed (biopsies) | 117
percentage of mean residual expression
  Tacrolimus dose | 0.676 [-1.159 to 2.511]
  Prednisone Dose | -1.687 [-3.27 to -0.104]
  Mycophenolate Mofetil Dose | -0.0035 [-0.013 to 0.006]
Statistical Analysis 1: Comparison: Lung Transplant Participants; P-value of tacrolimus dose; Test type: Other — Generalized estimating equation-adjusted linear models; p = 0.470, GEE-adjusted linear models
Statistical Analysis 2: Comparison: Lung Transplant Participants; P-value of Prednisone dose; Test type: Other — Generalized estimating equation-adjusted linear models; p = 0.037, GEE-adjusted linear models
Statistical Analysis 3: Comparison: Lung Transplant Participants; P-value of mycophenolate mofetil dose; Test type: Other — Generalized-estimating equation-adjusted linear models; p = 0.456, GEE-adjusted linear models

ADVERSE EVENTS:
Time Frame: from 1 month up to 18 months post-transplant
Arm/Group | Lung Transplant Participants
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

LIMITATIONS AND CAVEATS:
Higher than expected variance in MRE and missed study visits somewhat reduced statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT02278952/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT02278952/Prot_SAP_001.pdf